CLINICAL TRIAL: NCT06570213
Title: Evaluating The Efficacy Of Combined Cognitive Processing Therapy and Stellate Ganglion Blocks for PTSD: A Randomized Controlled Trial
Brief Title: Evaluating The Efficacy Of Combined Cognitive Processing Therapy and Stellate Ganglion Blocks for PTSD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Held, Research Director, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23091404
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Random assignment of eligible participants will occur in two steps using a custom computer randomization algorithm. First, participants will be randomly assigned to receive either two active SGB injections or two placebo saline injections. In the second stage of random assignment, participants will be randomly assigned to receive 1-week of CPT or daily symptom monitoring.
  As there will only be three treatment conditions of this study (SGB+CPT, SGB+Daily Monitoring, and Placebo Injection+CPT), individuals that are randomly assigned to the placebo injection group in the first stage of random assignment will automatically be assigned to receive CPT.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Stellate Ganglion Block + Cognitive Processing Therapy (Active Comparator): Participants in this arm will receive two active Stellate Ganglion Block Injections, two weeks apart. After receiving the first injection, participants will complete 10 sessions of Cognitive Processing Therapy over the course of one week.
  Interventions: Behavioral: Cognitive Processing Therapy; Drug: Stellate Ganglion Block
- Placebo Injection + Cognitive Processing Therapy (Sham Comparator): Participants in this arm will receive two placebo (saline) Injections, two weeks apart. After receiving the first injection, participants will complete 10 sessions of Cognitive Processing Therapy over the course of one week.
  Interventions: Behavioral: Cognitive Processing Therapy
- Active Stellate Ganglion Block + Daily Symptom Monitoring (Placebo Comparator): Participants in this arm will receive two active Stellate Ganglion Block Injections, two weeks apart. After receiving the first injection, participants will complete 5 sessions of daily symptom monitoring with a member of study staff over the course of one week.
  Interventions: Drug: Stellate Ganglion Block

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is a first-line, gold-standard psychotherapy intervention for the treatment of PTSD.
  Arms: Active Stellate Ganglion Block + Cognitive Processing Therapy; Placebo Injection + Cognitive Processing Therapy
Drug: Stellate Ganglion Block — Stellate Ganglion Blocks are an injection of local anesthetic into the stellate ganglion, a collection of nerves in the side of the neck.
  Arms: Active Stellate Ganglion Block + Cognitive Processing Therapy; Active Stellate Ganglion Block + Daily Symptom Monitoring

SUMMARY:
The purpose of this study is to understand if we can improve the treatment for posttraumatic stress disorder (PTSD). We are looking into whether the combination of Stellate Ganglion Block (SGB) treatment and Cognitive Processing Therapy (CPT) can reduce symptoms of PTSD. CPT is a trauma-focused talk therapy that can help identify and challenge unhelpful trauma-related beliefs about oneself, others, and the world. It is known to be a highly effective talk therapy for PTSD. SGB treatment is a procedure involving an injection of local anesthetic into a bundle of nerves located in the neck that is part of the sympathetic nervous system which controls our body's response to stressful situations and blocks pain.

The proposed project will systematically test whether combining CPT with SGB produces greater PTSD symptom reductions and functional improvements in the short- and longer-term up to 6-months follow-up compared to CPT (+Placebo) or SGB (+Daily Monitoring) alone.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Are fluent in English
* Have experienced a Criterion A traumatic event during their lifetime
* Have a PTSD diagnosis verified via the Clinician Administered PTSD Scale for DSM-5
* Have not previously received a Stellate Ganglion Block
* Have a smartphone that they can use for the entire duration of the study
* Are willing and able to receive 2 injections (SGB or placebo) 2 weeks apart at the Rush Pain Clinic
* Are willing and able to participate in daily Cognitive Processing Therapy or Daily Monitoring over the course of one week
* Are willing and able to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study

Exclusion Criteria:

* The traumatic event occurred in the past month
* They are currently suicidal or homicidal (i.e., plan and intent)
* They have unmanaged psychosis or mania
* They have not been on a stable dose of psychotropic medication for at least one month by the time of the baseline assessment or are planning to change their medications within 3 months of starting their participation in the study
* They have completed an evidence-based cognitive behavioral PTSD treatment (e.g., Cognitive Processing Therapy or Prolonged Exposure) in the past 3 months or are currently receiving an evidence-based PTSD treatment
* They have an intellectual disability or significant cognitive impairment that would prevent them from engaging fully in treatment
* They are currently on any blood-thinning medications or have a coagulopathy -They have any of the following conditions: a recent myocardial infarction, glaucoma, a pre- existing contralateral nerve palsy, severe emphysema, or a cardiac conduction blockade.
* They are allergic to any of the medications injected (i.e., ropivacaine, lidocaine, propofol)
* They have an active infection
* They have a serious or unstable medical illness or instability for which hospitalization may be likely within the next year
* They have a visual or auditory impairment that would prevent them from fully participating in study activities
* They are involved with current legal actions related to the traumatic event that is anticipated to be targeted during treatment
* They have substance dependence that, in the judgment of the Principal Investigator, may require hospitalization if substances were discontinued.
* Subjects who, at the time of consent, appear to have extenuating life circumstances (e.g., unstable housing, no internet access, etc.) which, in the judgment of the Principal Investigator, could affect the ability to deliver the intervention with fidelity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 | Baseline to 6 month follow up
  A clinician rated assessment of PTSD
PTSD Checklist for DSM-5 | Baseline to 6 month follow up
  A self-report measure of PTSD symptom severity

IPD SHARING:
Plan to Share IPD: No